CLINICAL TRIAL: NCT03298204
Title: A Multicenter Analysis of Definitive (Chemo)Radiotherapy With or Without Chemotherapy for Patients With Esophageal Cancer - 3JECROG-R01
Brief Title: Definitive (Chemo)Radiotherapy for Patients With Esophageal Cancer - 3JECROG R-01
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Hebei Medical University Fourth Hospital (Other); Fujian Cancer Hospital (Other Government); Anyang Tumor Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Affiliated Hospital of Hebei University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Beijing Hospital (Other Government); Tengzhou Central People's Hospital (Other Government); PLA Army General Hospital (Unknown)
Responsible Party: Principal Investigator, Zefen Xiao, MD, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: 3JECROG R-01
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Esophagus Cancer; Chemoradiation; Chemotherapy Effect; Radiotherapy Side Effect
MeSH Terms: conditions — Esophageal Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chemoradiotherapy
- Chemoradiotherapy following chemotherapy
- Chemoradiotherapy followed by chemotherapy

SUMMARY:
The aim of this observational study is to retrospectively collect survival data for 3000 primary esophageal cancer patients from multicenter between January 2000 to present. Based on a Cox model, we want to develope a nomogram that predicts local recurrence, distant metastases, and survival for patients treated with radiotherapy or chemoradiotherapy with or without chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma, adenocarcinoma of the esophageal or esophagogastric junction Unresectable or potentially resectable tumor (cT3-4N0-1M0-M1b, without visceral metastasis, according to AJCC 6th) based on standard primary staging by EUS and CT
* Age>18 years
* No distant metastasis other than supraclavicular lymph nodes
* No prior history of thoracic radiation
* Patients must have normal organ and marrow function as defined below: Leukocytes: greater than or equal to 3,500 G/L; Platelets: greater than or equal to 100,000/mm3 .Hemoglobin:greater than or equal to 10g/L .Total bilirubin: within normal institutional limits; AST/ALT: less than or equal to 1.5 times the upper limit; Creatinine within normal upper limits

Exclusion Criteria:

* Patients with other cancer history except cervical carcinoma in situ and non-malignant melanoma skin cancer during 5 years before diagnosis of esophageal cancer
* Pregnant or lactating females
* Contraindication for radiotherapy or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal or esophagogastric junction cancer
Sampling Method: Probability Sample
Enrollment: 2762 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year
Overall survival | 2 year

SECONDARY OUTCOMES:
Progress free survival | 1 year
Progress free survival | 2 year
Locoregional recurrence free survival | 1 year
Locoregional recurrence free survival | 2 year
Distant metastasis free survival | 1 year
Distant metastasis free survival | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, National Cancer Center, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, China